CLINICAL TRIAL: NCT03830385
Title: Open-Label, Multicenter, Phase Ⅱ Study Of Paclitaxel (Albumin Bound),Bleomycin And Cisplatin Or Carboplatin As First-Line Treatment In Patients With Recurrent Or Metastatic Squamous Cell Carcinoma Of The Head And Neck
Brief Title: Paclitaxel (Albumin Bound),Bleomycin And Cisplatin Or Carboplatin for Recurrent Or Metastatic Squamous Cell Carcinoma Of The Head And Neck
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-138
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Squamous Cell Carcinoma Of The Head And Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel (Albumin Bound),Bleomycin and Cisplatin or (Experimental)
  Interventions: Drug: PaclitaxelPaclitaxel (Albumin Bound),Bleomycin combined with Cisplatin or Carboplatin

INTERVENTIONS:
Drug: PaclitaxelPaclitaxel (Albumin Bound),Bleomycin combined with Cisplatin or Carboplatin — All patients enrolled in the study will accept Paclitaxel (Albumin Bound),Bleomycin combined with Cisplatin or Carboplatin as their firstline chemotherapy

SUMMARY:
The purpose of this single arm, phase Ⅱ clinical trail is to determine the safety and efficacy of paclitaxel (albumin bound),bleomycin and cisplatin or carboplatin in the treatment of recurrent Or metastatic squamous cell carcinoma of the head and neck

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved squamous cell carcinoma of the head and neck;
* stage IVc according to Union for International Cancer Control (UICC) edition VIII, or recurrent disease after chemotherapy and/or radiotherapy;
* 18 years or older; without other malignancy;
* proper functioning of the major organs.

Exclusion Criteria:

* allergic to paclitaxel (albumin bound) or bleomycin or cisplatin or carboplatin ;
* female within gestation period or lactation;
* patients received drug of other clinical trial within 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China